CLINICAL TRIAL: NCT03315637
Title: Fetal Endoscopic Surgery for Spina Bifida
Acronym: FESSB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR(AMI)152/2015
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Neural Tube Defects; Spina Bifida, Open; Myelomeningocele; Fetal Disease; Hydrocephalus; Chiari Malformation Type 2; Congenital Abnormality; Surgery; Maternal, Uterus or Pelvic Organs, Affecting Fetus
MeSH Terms: conditions — Neural Tube Defects; Spina Bifida Cystica; Meningomyelocele; Fetal Diseases; Hydrocephalus; Arnold-Chiari Malformation; Congenital Abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetoscopic repair of spina bifida (Experimental): This is a single arm study, all patients will receive a fetoscopic repair of the spina bifida
  Interventions: Procedure: Fetoscopic repair of spina bifida

INTERVENTIONS:
Procedure: Fetoscopic repair of spina bifida — Fetoscopic intrauterine repair of open spina bifida

SUMMARY:
This study aims to assess the feasibility to perform a fetoscopic prenatal repair of an open neural tube defect, and secondly to assess the maternal, fetal and neonatal outcomes.

DETAILED DESCRIPTION:
Introduction:

Spina bifida is a congenital malformation characterized by a failure in neural tube closure. Unprotected fetal neural tissue at the spine level undergoes not only progressive neurodegeneration in spinal cord, but also the impairment in brain development, hindbrain herniation or Chiari II malformation probably due to pressure disturbances resulting from a continuous leakage of cerebrospinal fluid through the defect. The neurological consequences at birth are irreversible and sometimes devastating, including paraplegia, sphincter urinary and fecal incontinence, hydrocephalus, cranial nerve disturbances, respiratory problems and death due to spinal cord injury and brain maldevelopment.

Intrauterine fetal open repair of the defect has proved to improve hindbrain herniation and decrease the need of cerebrospinal shunting.

Hypothesis:

The investigators hypothesize that minimally invasive surgery of spina bifida is feasible and may minimize surgical aggression and obstetrical complications, with similar neonatal and neurological results.

Intervention:

In this study the investigators propose a fetoscopic skin closure technique. After a maternal laparotomy the uterus is exteriorized, the amniotic cavity is accessed by fetoscopic approach. The placode is dissected from the surrounding tissue and dropped into the opened spinal canal, untethered. Part of the cystic tissue is resected. The edges are then closed to the midline.

Follow up:

After surgery patients are followed up at the Fetal Medicine Unit every one or two weeks.

The mode of delivery is decided according to obstetric criteria. Neonates will be examined at birth, and followed up regularly at least until 30 months. Patients are lifetime followed up by our Multidisciplinary myelomeningocele (MMC) Committee that comprises professionals from the Spina Bifida Unit, Neonatologists, Pediatric Surgeons, Pediatric Urologist, Pediatric Orthopedic Surgeons, Radiologists, Rehabilitation, Pathologists, Pediatric Neurosurgeons, Obstetricians and Fetal Therapists.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18 years old
* Singleton pregnancy
* Gestational age between 18 0/7 weeks and 26 6/7 weeks
* Isolated neural tube defect between T1 and S1
* Cerebellar herniation (Chiari type II)

Exclusion Criteria:

* Fetal anomalies non related to neural tube defect (NTD) including chromosomal abnormalities
* Body mass index > 35 kg/m2
* Maternal disorders contraindicating surgery
* Genetic anomalies with poor prognosis
* Sever kyphosis (>30º)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Capability to achieve successful closure of the neural tube defect by fetoscopic surgery (yes/no) | Time of procedure (day 0)
  Binary variable (yes/no) describing if the neural tube defect has been successfully closed, (placode dissected and dropped into the open spinal canal, cystic tissue resected and edges closed to the midline), by fetoscopic surgery, and without conversion to open surgery

SECONDARY OUTCOMES:
Operating time (minutes) | Time of procedure (day 0)
  Time between the skin opening and skin closure
Fetoscopy time (minutes) | Time of procedure (day 0)
  Time between the introduction of the first cannula and the removal of the last cannula
Hospital stay (days) | Between procedure and delivery, up to 21 weeks
  Time between hospital admission and discharge

OTHER OUTCOMES:
Post-operative hemoglobin (g/dL) | 24 hours after procedure
  Hemoglobin level after the procedure
Blood transfusion (yes/no) | Between procedure and discharge, up to 21 weeks
  Binary variable describing if a transfusion of blood derivates is carried out between the time of procedure and discharge
Gestational age at delivery (weeks and days as x/7) | At birth, up to 21 weeks after procedure
  Gestational age at birth
Surgery to delivery interval (days) | At birth, up to 21 weeks after procedure
  Interval between surgery and birth
Premature rupture of membranes (PROM) (yes/no) | Between the procedure and 37 weeks of pregnancy (18 weeks after procedure)
  Binary variable describing amniotic fluid leakage before the onset of labor
Chorioamnionitis (yes/no) | Between the procedure and birth, up to 21 weeks after procedure
  Binary variable describing the presence of a chorioamnionitis between the procedure and birth
Oligohydramnios without PROM (yes/no) | Between the procedure and birth, up to 21 weeks after procedure
  Binary variable describing the presence of a oligohydramnios (deepest pool < 2 cm) without evidence of vaginal amniotic fluid leakage
Placental abruption (yes/no) | Between the procedure and birth, up to 21 weeks after procedure
  Binary variable describing the presence of a placental abruption
Mode of delivery (vaginal / cesarean) | At birth, up to 21 weeks after procedure
  Binary variable describing the mode of delivery, vaginal or cesarean section
Uterine dehiscence (yes/no) | At birth, up to 21 weeks after procedure
  Binary variable describing the presence of a uterine dehiscence, regardless of whether it is symptomatic or it is diagnosed at the time of cesarean section
Acute Pulmonary edema (yes/no) | Between the procedure and birth, up to 21 weeks after procedure
  Binary variable describing the presence of a maternal pulmonary edema, regardless of the severity, between the procedure and discharge.
Closure of the spinal defect (yes/no) | Between birth and 1 month of life
  Binary variable describing the watertight closure of the defect
Maintenance of the neurological level (Better / same / worse) | 1 month of life
  Categorical variable describing if the postnatally assessed neurological level is better / same or worse than the level assessed prenatally before the procedure. It will be assessed by physical examination
Reversal of Chiari malformation(completely reversed / mild improvement / no improvement) by MRI | 1 month of life
  Categorical variable comparing the postnatal and prenatal MRI assessment of the Chiari malformation
Ventriculoperitoneal shunting (yes/no) | Between birth and 12 months
  Binary variable describing the need of a ventriculoperitoneal shunting

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Maroto A, Illescas T, Melendez M, Arevalo S, Rodo C, Peiro JL, Belfort M, Cuxart A, Carreras E. Ultrasound functional evaluation of fetuses with myelomeningocele: study of the interpretation of results. J Matern Fetal Neonatal Med. 2017 Oct;30(19):2301-2305. doi: 10.1080/14767058.2016.1247262. Epub 2017 Jan 16. PMID 27997256
- [Background] Belfort MA, Whitehead WE, Shamshirsaz AA, Bateni ZH, Olutoye OO, Olutoye OA, Mann DG, Espinoza J, Williams E, Lee TC, Keswani SG, Ayres N, Cassady CI, Mehollin-Ray AR, Sanz Cortes M, Carreras E, Peiro JL, Ruano R, Cass DL. Fetoscopic Open Neural Tube Defect Repair: Development and Refinement of a Two-Port, Carbon Dioxide Insufflation Technique. Obstet Gynecol. 2017 Apr;129(4):734-743. doi: 10.1097/AOG.0000000000001941. PMID 28277363